CLINICAL TRIAL: NCT06003504
Title: The Impact of First Aid Training, Delivered Via a Face-to-face or Blended Learning Approach, on Learning Outcomes and Helping Behaviour of Adult Laypeople in Rwanda: a Randomised Controlled Trial
Brief Title: The Impact of First Aid Blended Learning Training on Learning Outcomes and Helping Behaviour of Adult Laypeople in Rwanda
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Evidence-Based Practice, Belgium (Other)
Collaborators: Rwanda Red Cross (Unknown); Belgian Red Cross (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: FABL-001
Record Dates: First submitted 2023-08-15; First posted 2023-08-22 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Emergencies; Injuries; Illness Physical
Keywords: First aid; Blended learning; Laypeople
MeSH Terms: conditions — Emergencies; Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: This is a randomised controlled trial in which the allocation is done at the level of the individual participant.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- First aid training with blended learning approach (Experimental): Participants follow a first aid training delivered through a blended learning approach.
  Interventions: Other: First aid training with blended learning approach
- First aid training with face-to-face approach (Active Comparator): Participants follow a first aid training delivered through a conventional face-to-face approach.
  Interventions: Other: First aid training with face-to-face approach
- Waitlist control (No Intervention): Participants do not receive any training

INTERVENTIONS:
Other: First aid training with blended learning approach — The content of the first aid blended learning training is standardised and based on the 2021 edition of the Basic First Aid in Africa manual from the Belgian Red Cross, covering first aid general principles and instructions for:
  * emergencies (i.e. choking, unconsciousness with and without normal breathing, chest discomfort and stroke, poisoning, and severe external bleeding);
  * injuries (i.e. skin wounds, burns, and injuries to muscles, joints, limbs, head, neck, and back);
  * illnesses (i.e. fainting, fever, fits, and diarrhoea).
  The training consists of 2 consecutive parts:
  1. First aid theory is learned independently in a mobile application followed by an online test to ob-tain an admission ticket for the subsequent in-class training;
  2. First aid skills are practiced during a 1-day in-class training facilitated by a certified first aid instructor of the Rwanda Red Cross.
  Participants get at least 10 days to learn in the mobile application and obtain the admission ticket.
  Other Names: First Aid Blended Learning (FABL)
  Arms: First aid training with blended learning approach
Other: First aid training with face-to-face approach — The content of the first aid face-to-face training is standardised and based on the 2021 edition of the Basic First Aid in Africa manual from the Belgian Red Cross, covering first aid general principles and instructions for:
  * emergencies (i.e. choking, unconsciousness with and without normal breathing, chest discomfort and stroke, poisoning, and severe external bleeding);
  * injuries (i.e. skin wounds, burns, and injuries to muscles, joints, limbs, head, neck, and back);
  * illnesses (i.e. fainting, fever, fits, and diarrhoea).
  The training consists of a 3-days in-class training with lectures and practical exercises on first aid the-ory and skills, facilitated by a certified first aid instructor of the Rwanda Red Cross.
  Other Names: Basic First Aid in Africa (BFA)
  Arms: First aid training with face-to-face approach

SUMMARY:
The goal of this study is to assess the impact of a first aid training delivered through a blended learning approach on learning outcomes and helping behaviour in adult laypeople in Rwanda.

Participants will be randomly assigned to either:

* a first aid training with blended learning approach;
* a first aid training with conventional face-to-face approach;
* no first aid training.

All participants will be asked before, immediately after, and 6 months after the first aid trainings to complete

* a questionnaire on first aid-related knowledge, self-efficacy, and willingness to help;
* a practical test on first aid-related skills.

The helping behaviour of the participants will be surveyed before and 6 months after the first aid trainings have been completed.

Researchers will compare the effects in learning outcomes and helping behaviour after 6 months between:

* the first aid training with blended learning approach and no first aid training;
* the first aid training with blended learning approach and first aid training with conventional face-to-face approach.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥ 18 years) laypeople
* Access to a smartphone or tablet, which is able to install and run a mobile application

Exclusion Criteria:

* Having attended a first aid training in the past
* Having an academic or professional background in the (para)medical field

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 540 (Actual)
Dates: Start 2023-07-13 (Actual); Primary Completion 2024-03-24 (Actual); Study Completion 2024-03-24 (Actual)

PRIMARY OUTCOMES:
First aid knowledge | Before, immediately after, and 6 months after the first aid trainings
  20-item multiple choice questionnaire about first aid topics using a numerical scale. Possible scores range from 0 to 20, with higher scores meaning a better outcome.

SECONDARY OUTCOMES:
First aid skills | Before, immediately after, and 6 months after the first aid trainings
  22-item observation checklist about first aid practical skills using a numerical scale. Possible scores range from 0 to 30, with higher scores meaning a better outcome.
First aid self-efficacy | Before, immediately after, and 6 months after the first aid trainings
  10-item scenario-based questionnaire using a 5-point Likert scale assessing self-efficacy concerning first aid topics. Possible scores range from 0 to 40, with higher scores meaning a better outcome.
First aid willingness to help | Before, immediately after, and 6 months after the first aid trainings
  6-item scenario-based questionnaire using a 5-point Likert scale assessing willingness to help concerning first aid topics. Possible scores range from 0 to 24, with higher scores meaning a better outcome.
Helping behaviour in the past 6 months | Before and 6 months after the first aid trainings
  Structured questionnaire to survey the helping behaviour and to gauge the potential barriers and facilitators.

OTHER OUTCOMES:
Costs | Before, immediately after, and 6 months after the first aid trainings
  Costs associated with a first aid training, relatively to the gain in knowledge.

CONTACTS AND LOCATIONS:
Overall Officials: Emmy De Buck, PhD, Principal Investigator — Centre for Evidence-Based Practice, Belgium
Locations (1):
- Rwanda Red Cross, Kigali, Rwanda

IPD SHARING:
Plan to Share IPD: Undecided